CLINICAL TRIAL: NCT04710446
Title: Clinical Characteristics, Treatments, and Outcomes of MI Patients Presenting With Normal ECG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Normal MI
Record Dates: First submitted 2020-12-02; First posted 2021-01-14 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Non-ST Elevated Myocardial Infarction; Electrocardiography
Keywords: Clinical Characteristics; Treatments; Outcomes; normal ECG
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- NSTEMI Patients presenting with normal ECG: NSTEMI Patients presenting with normal ECG
- NSTEMI Patients presenting with isolated T wave inversion: NSTEMI Patients presenting with isolated T wave inversion
- NSTEMI Patients presenting with transient ST-segment elevation: NSTEMI Patients presenting with transient ST-segment elevation
- NSTEMI Patients presenting with resting U wave inversion: NSTEMI Patients presenting with resting U wave inversion
- NSTEMI Patients presenting with low QRS voltage: NSTEMI Patients presenting with low QRS voltage

SUMMARY:
the investigators aimed to analyzed data for hospitalized MI patients with normal ECG.

DETAILED DESCRIPTION:
The electrocardiogram (ECG) at presentation is a useful tool for risk prediction. Patients with ACS（Acute Coronary Syndromes） and ST-segment depression on ECG have a worse prognosis than patients with a normal ECG. ST-segment depression is not only a qualitative marker, but also a quantitative marker of risk, because the number of leads with ST-segment depression and the magnitude of ST-segment depression (either within a single lead or as sum over all leads) are indicative of the extent of ischaemia and correlate with prognosis.The presence of ST-segment depression >1 mm in >_6 leads in conjunction with ST-segment elevation in aVR and/or V1, particularly if the patient presents with haemodynamic compromise, suggests multivessel ischaemia or severe left main coronary artery stenosis. However,in patients presenting without persistent ST-segment elevation,the clinical features, treatments, and outcomes in patients with normal ECG is still unclear.

ELIGIBILITY:
Inclusion Criteria:all patients hospitalized with a principal diagnosis of non-ST-segment elevation infarction (NSTEMI) according to the current ACC/AHA guidelines.

exclusion criteria: end-stage organic disease, thrombotic hematological disorders, and poor echogenicity

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSTEMI Patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
MACE within 2 weeks | within 2 weeks
  Major Adverse Cardiovascular Events within2 weeks
MACE within 1 year | within 1 year
  Major Adverse Cardiovascular Events in-hospital within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: yansheng Huang, Study Director — Henan Provincial People's Hospital
Locations (1):
- Henan province people's hospital, Zhengzhou, Henan, China